CLINICAL TRIAL: NCT06291506
Title: : SUbstrate Ablation in Persistent Atrial Fibrillation for Elimination of Recurrences (SUPAFER): a Multicentre Randomized Clinical Trial to Assess Pulmonary Vein Isolation Alone or Combined With Linear Ablation.
Brief Title: SUbstrate Ablation in Persistent Atrial Fibrillation for Elimination of Recurrences (SUPAFER).
Acronym: SUPAFER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario La Paz (Other)
Responsible Party: Principal Investigator, Dr. Sergio Castrejón-Castrejón, Consultant of Cardiology, main coinvestigator, coordinator., Hospital Universitario La Paz
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 6270
Record Dates: First submitted 2024-01-08; First posted 2024-03-04 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Persistent and Long Lasting or Chronic Atrial Fibrillation; Atrial Fibrillation Ablation; Linear Left Atrial Ablation; Daily Transtelephonic Electrocardiogram

STUDY DESIGN:
Intervention Model Description: 1:1 randomization
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pulmonary veins isolation plus linear left atrial ablation. (Experimental)
  Interventions: Other: Radiofrequency ablation of heart atrial tissue.
- Pumonary veins isolation only. (Active Comparator)
  Interventions: Other: Radiofrequency ablation of heart atrial tissue.

INTERVENTIONS:
Other: Radiofrequency ablation of heart atrial tissue. — Ablation with radiofrequency, advances techniques: contact force-guided, improved tissue temperature sensors, automark algorithms.

SUMMARY:
Antecedents: electrical isolation of pulmonary veins is the standard treatment for patients with atrial fibrillation. However, its efficacy is lower in persistent and chronic forms of this arrhythmia compared to paroxysmal atrial fibrillation. Many complementary techniques have been proposed, that added to pulmonary veins isolation, may reduce the recurrence rate of atrial fibrillation. However, none of them has obtained consistent results. Linear ablation aims to parcellate and modify the left atrial substrate responsible for atrial fibrillation maintenance. Previous studies have offered contradictory results using linear ablation.

Methods: SUPAFER is a multicenter, 1:1 randomized clinical trial that compares the efficacy of pulmonary veins isolation alone vs pulmonary vein isolation plus an specific protocol of left atrial linear ablation. Contrary to previous studies, the specific SUPAFER linear ablation is systematic, homogeneous and target atrial areas that have not been systematically ablated in previous trials. The trial aims at demonstrating the superiority of the combined ablative approach during 1-year follow-up. Daily transtelephonic ECG samples a 30 days continuous ECG monitoring are used to maximize de detection of recurrences, even asymptomatic.

ELIGIBILITY:
Inclusion Criteria:

* Persistent atrial fibrillation documented with electrocardiogram and defined as: persistent (continuous AF duration >1 week) or long-lasting persistent (continuous AF duración >1 year).
* One of the following additional criteria: 1)symptomatic AF, 2)recurrence despite antiarrhythmic drugs or after electrical cardioversion, 3)tachymiopathy, 4)heart failure, 5)antiarrhythmic drugs either not tolerated or rejected or considered inadequate by the patient or an electrophysiology specialist, 6)preference for ablation explicitly manifested by the patient.
* Age >=18 years and written informed consent.

Exclusion Criteria:

* AF with a reversible cause.
* Previous pulmonary veins isolation or left atrial linear ablation.
* Cardiac surgery, acute coronary syndrome, percutaneous coronary intervention o ischaemic stroke <1 month before ablation.
* Intracranial haemorrhage <3 months before ablation.
* Ablation contraindicated due to 1)absolute contraindication for oral anticoagulants, 2)persistent atrial thrombus, 3)pregnancy, 4)extreme fragility and 5)life expectancy <1 year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Recurrences of sustained >30 secons atrial arrhythmias measured by daily ECG samples (Kardia Alivecor) and 30 days continuous Holter. | through study completion, 1 year follow-up
  Atrial fibrillation, atrial tachycardia (atrial flutter).

SECONDARY OUTCOMES:
Acute intraprocedure efficacy. | during the ablation procedure and up to 2 months blanking perior
  Rate of: AF termination to sinus rhythm, organization to atrial tachycardia and non inducibility of AF or atrial tachycardia.
Complications. | through study completion, 1year follow-up
  Complications associated to the ablation procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- La Paz University Hospital - IdiPaz, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No